CLINICAL TRIAL: NCT05551286
Title: The 'Young Adult Taking Action' Programme for Young Adult Cancer Survivors: a Feasibility Study Evaluating Content and Delivery
Brief Title: Feasibility of the YATAC Programme
Acronym: YATAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1234
Record Dates: First submitted 2022-09-08; First posted 2022-09-22 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Rehabilitation; Young adults
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Young Adults Taking Action (Experimental): The programme is person-centered, goal-oriented, and peer-based and is structured around a 5-day residential stay, an online follow-up after five weeks and a 2-day residential follow-up stay after ten weeks.
  Interventions: Other: A rehabilition programme for young adult cancer survivors

INTERVENTIONS:
Other: A rehabilition programme for young adult cancer survivors — The programme consists of 22 sessions focusing on; 1) everyday life (energy conservation, cognitive challenges, fatigue); 2) Physical activity; 3) psychological issues; 4) work and study d; 5) sexuality and relationship; 7) rights and finance, and 8) goal setting. The sessions include both education, workshops, and engagement in different activities and will be delivered by a multidisciplinary team.

SUMMARY:
Young adult cancer survivors (YACS) aged 18-39 report physical and psychosocial late effects following cancer treatment, impairing quality of life and participation in everyday life. To address such multifactorial challenges complex or multicomponent rehabilitation interventions are needed. Based on this, the 'Young Adult Taking Action' (YATAC) programme was developed to increase participation in everyday life and improve health-related quality of life. The development of the intervention is guided by the British Medical Research Council's guidance (MRC) and the framework for the co-production and prototyping of public health interventions by Hawkins et al.

The present study will investigate the acceptability and fidelity of the intervention at the research clinic of REHPA, the Danish Knowledge Centre for Rehabilitation and Palliative Care in Nyborg, Denmark. A mixed method one-armed feasibility study will be conducted and the results of the study will be used to revise version 1.0 of the programme.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-39 years old at baseline
* Have had any type of cancer
* Have completed primary/active cancer directed treatment (cytotoxic chemotherapy, radiation therapy and/or definitive surgical intervention, while current hormonal treatments or maintenance therapies are permissible)
* Determined a need for rehabilitation determined by the REHPA scale (a linear analogue scale, where the participants indicate how close they are to living the life they desire after ending cancer treatment). The scale ranges from 0= 'goal reached' to 9= 'infinitely far from'
* Have access to a device with Internet options (i.e., smartphone or tablet)

Exclusion Criteria:

* Dependent in basic personal activities of daily living (personal care, dressing and eating)
* No permanent residence in Denmark
* Not able to speak and understand Danish

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Acceptability; Affective attitude | 10 weeks
  The participants feelings about the intervention. Scores between 0-5, with higher scores indicating better feeling.
Fidelity | 10 weeks
  Defined as the consistency of whether the intervention was implemented as intended. The professionals register to what extent they have implemented the session as intended on a 5-point Likert scale. Scores between 0-5, with higher scores indicating higher consistency.
Dose | 10 weeks
  Defined as the quantity of intervention implemented. The professionals will report the number of elements implemented and the time used. In addition, the professional will give information on reasons for deviation from the manual.
Adaptions | 10 weeks
  Defined as any adjustments made to the intervention. The professionals register and describe any adaptions they make and the reasons for this.
Acceptability; burden | 10 weeks
  The participants perceived amount of effort required to participate. Scores between 0-5, with higher scores indicating high degree of effort.
Acceptability; Ethicality | 10 weeks
  The participants opinion about the intervention's fit with their individuals value system. Scores between 0-5, with higher scores indicating higher consistency with value system.
Acceptability; intervention cohesion | 10 weeks
  The participants understanding of the intervention and how it works. Scores between 0-5, with higher scores indicating higher understanding of the intervention.
Acceptability; opportunity costs | 10 weeks
  The participants experience of opportunity costs, like benefits, values, or profits that must be given up to engage in the intervention. Scores between 0-5, with higher scores indicating higher degree of giving up on opportunity costs, like benefits, values, or profits.
Acceptability; Perceived effectiveness | 10 weeks
  The participants experience of perceived effectiveness of the intervention. Scores between 0-5, with higher scores indicating higher degree of perceived effectiveness of the intervention.
Acceptability; Self-efficacy | 10 weeks
  The participants confidence that they can perform the behavior(s) required to participate in the intervention. Scores between 0-5, with higher scores indicating higher confidence that they can perform the behavior(s) required to participate in the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Aagesen, PhD student, Principal Investigator — The University of Southern Denmark
Locations (1):
- REHPA, The Danish Knowledge Centre for Rehabilitation and Palliative Care, Nyborg, The Region of Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No